CLINICAL TRIAL: NCT07000279
Title: Assessment of Feasibility, Functionality and Usability of an Hybrid Assistive Exoskeleton for Upper Limb: a Pilot Study
Brief Title: Assessment of Feasibility, Functionality and Usability of an Hybrid Assistive Exoskeleton for Upper Limb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Collaborators: Università Campus Bio-Medico di Roma (UCBM) (Unknown); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Principal Investigator, Emanuele Gruppioni, Engineer, Orthopaedic Technician, Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-PAI-03-23
Record Dates: First submitted 2025-05-12; First posted 2025-06-02 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Upper Limb Deficits
Keywords: assistive exoskeleton; upper arm; post stroke; brachial plexus injury; orthesis; functional electrical stimulation; activity of daily living; portable device
MeSH Terms: interventions — Activities of Daily Living; Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruited subjects with exoskeleton (Experimental): Subjects are asked to perform the study procedure while wearing the assistive device
  Interventions: Device: Assistive exoskeleton for activities of daily living (ADLs); Device: Assistive exoskeleton for box and block; Device: Assistive exoskeleton for maximum reaching height
- Recruited subjects without exoskeleton (No Intervention): Subjects are asked to perform the study procedure not wearing the assistive device

INTERVENTIONS:
Device: Assistive exoskeleton for activities of daily living (ADLs) — Portable assistive exoskeleton to support upper limb movement during activities of daily living
  Arms: Recruited subjects with exoskeleton
Device: Assistive exoskeleton for box and block — Portable assistive exoskeleton to support box and block test execution
  Arms: Recruited subjects with exoskeleton
Device: Assistive exoskeleton for maximum reaching height — Portable assistive exoskeleton to raise the upper limb at the maximum of its capability to reach objects at different heights
  Arms: Recruited subjects with exoskeleton

SUMMARY:
People affected by stroke or brachial plexus injuries experience huge impairment in using upper limbs for everyday life activities. Brachial plexus is responsible of sensory-motor innervation of the whole upper limb, the shoulder and also a part of the chest. The majority of such injuries is caused by traumatic events that involve young and healty people in most cases and motor impairment varies together with either the type (complete or incomplete) or the site of injury. It follows the need to realize devices capable of restoring people everyday life independence.

To assist these patients, the most common solutions are passive ortheses that give support to shoulder and forearm without actively enhancing limb functionalities. MyoPro (by MIT, Myomo1) is the only active device available for elbow and wrist, even not completely proven for everyday life yet. It comes from scientific evidences that gravity compensation and functional electrical stimulation (FES) are considerable techniques for rehabilitation of brachial plexus injuries and post-stroke patients. According to the most recent results, hybrid systems that combine FES with robotic joints seem to give interesting benefits in such the contexts taken into account.

The goal of this clinical trial is to assess feasibility, functionality and usability of a new assistive, hybrid, active and portable orthesis for upper limb aimed at improving motor functionality of brachial plexus injuries patients. Complying with weight and size requirements, the device under investigation is designed to assist the whole upper limb with its two modules: a robotic exoskeleton to actively give assistance to shoulder and elbow and a FES module to assist wrist and hand.

The main points the clinical trial aims to address concern:

* number and type of adverse events (device failures and malfunctioning, subjects injuries) during use
* evaluation of change in performance with and without the device
* usability and satisfaction after use
* effectiveness

Post-stroke and brachial plexus injuries patients (with Medical Research Council Scale for Muscle Strength equal to or more than 2) will be enrolled and asked to perform the following tasks with and without wearing the device:

* box and block test
* vertical reaching
* activities of daily living (ADLs) such as eating and drinking

Study procedure consists of 6 session outlined as follows:

* Session 1: enrollment
* Session 2: tuning and familiarization with device modules
* Session 3: tasks execution and outcomes measurement
* Session 4: tasks execution and outcomes measurement
* Session 5: tasks execution and outcomes measurement
* Session 6: extra session for any tasks from sessions 3,4,5 which required further investigations Each session will last 90 minutes at most. A preliminary phase will envolve healthy subjects that will be asked to perform the same tasks listed above. These tests will be useful to evaluate performances, functionalities and effectiveness of the modular solutions adopted, to improve the user experience of the device and to finalise the experimental procedure to follow with patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* post-stroke or brachial plexus injuries patients
* upper limb motor deficit patients with Medical Research Council (MRC) Scale for Muscle Strength equal to or more than 2
* number of months after lesion higher than 6
* cognitive ability to follow instruction
* no Functional Electrical Stimulation (FES) treatment within 6 months prior to the enrollment
* absence of communication deficit

Exclusion Criteria:

* other nuerological or orthopaedic impairments
* pain in injuried upper limb (Numeric Rating Scale (NRS) higher than 4)
* cognitive impairments (Mini-Mental State Examination (MMSE) lower than 24)
* implantable devices that can interfere with FES
* muscle/neurological diseases that can get worse with FES
* fever or infection
* pregnancy or breastfeeding
* absence of patient informed consent in written form
* unstable medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events occurred during use of the exoskeleton | During the intervention at days 2, 3, 4, 5
  Number of device failures and malfunctioning, device-related harms during device use
Change of score in Box and Blocks Test | During the intervention at days 3, 4, 5
  The box and block test measures how many cubic wooden blocks the subject is able to move from one side of a wooden box to the other side in 60 seconds. The subject is asked to perform the Box And Blocks test while wearing the device and without the device for comparison.
Change in performance during the execution of activities of daily living (ADLs) | During the intervention at days 3, 4, 5
  The subject is asked to perform different ADLs while wearing the device and without the device. Time for the execution and successful rate of activities are registered for comparison.
Change in kinematics during execution of tasks | During the intervention at days 3, 4, 5
  The subject is asked to perform the box and block test, maximum reaching height task and activites of daily living while wearing the device in assitive mode and without the device. The experimental setup is provided with Magneto-Inertial Measurement Unit (M-IMU) sensors capable to measure speed and smoothness of movements in both cases for comparison.
Change in upper limbs muscles activation during execution of tasks | During the intervention at days 3, 4, 5
  The subject is asked to perform the box and block test, maximum reaching height task and activites of daily living while wearing the device in assitive mode and without the device. The experimental setup is provided with surface EMG sensors capable to measure upper limb muscles activation in both cases for comparison.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | During the intervention at days 3, 4, 5
  SUS is a questionnaire aiming at measuring the perceived usability of the device. It's a 10-item questionnaire, 5-points Likert scale with item score ranging from 1 (strongly disagree) to 5 (strongly agree). In SUS score calculation, each item's score contribution will range from 0 to 4 with the final score obtained by summing the score contributions from each item and multiplying it by 2.5, in order to have a value in the range of 0 to 100. The higer the final score, the better the outcome.
Quebec User Evaluation of Satisfaction with assistive Technology questionnaire (QUEST) | During the intervention at days 3, 4, 5
  QUEST is a questionnaire aiming at measuring the perceived satisfaction of the device after use. It's a 12-item questionnaire, with item score ranging from 1 (worst) to 5 (best). The final score is obtained as an average of the items scores. The higer the final score, the better the outcome.
Numeric Rating Scale (NRS) for satisfaction | During the intervention at days 3, 4, 5
  A custom NRS 0-10 is created to measure the perceived level of acceptance of the device after use. The subject is asked to evaluate its perception of weight, comfort, safety and assistance wearing the device, with item score ranging from 0 (best) to 10 (worst). The higher the scores, the worse the outcome.
Numeric Rating Scale (NRS) for pain evaluation | During the intervention at days 3, 4, 5
  The subject is asked to evaluate its level of musculoskeletal pain after use with a score ranging from 0 (no pain) to 10 (max pain). The higher the score, the worse the outcome.
NASA Task Load Index (NASA-TLX) | During the intervention at days 3, 4, 5
  NASA-TLX is used with the aim of measuring the effectiveness of the device after use. It is a multi-dimensional rating procedure that provides an overall workload score based on a weighted average of ratings on six subscales: Mental Demands, Physical Demands, Temporal Demands, Own Performance, Effort, and Frustration. For each task or group of tasks, the subject is asked to select an option for each of the 15 comparison cards given (to obtain weights) and to express a score ranging from 1 (low/good) to 20 (high/poor) for each subscale (rate). The final workload score is computed by multiplying each rating by the weight given to that factor by that subject, then the sum of the weighted ratings for each task is divided by 15. The higer the final score, the worse the outcome.
Flow State Scale (FSS) | During the intervention at days 3, 4, 5
  FSS is a questionnaire aiming at measuring the user experience of the device during use. It's a 36-item questionnaire, with item score ranging from 1 (strongly disagree) to 5 (strongly agree). As 5-point Likert scale with 4 items per 9 subscales, the item scores for each dimension are summed and then divided by four, to obtain flow dimension item-average scores. The higer the final score, the better the outcome.
Category-Ratio 0-10 scale (Borg CR-10) | During the intervention at days 3, 4, 5
  Borg CR-10 Scale is a subjective measure of perceived exertion or intensity during the execution of tasks. Body sensations under evaluation concern heart rate, breath rate and muscle fatigue with item score ranging from 0 (nothing at all) to 10 (maximum). The higher the single scores, the worse the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Protesi Inail, Budrio, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Demographic and clinical data collected during the trial will be anonymized and aggregated prior to sharing
Time Frame: Within one year after trial conclusion (december 2025)
Access Criteria: Anonymized not aggregated data could be available upon request

REFERENCES:
- [Background] A. M. Stewart, C. G. Pretty, M. Adams, and X. Chen, "Review of Upper Limb Hybrid Exoskeletons," IFAC-Pap., vol. 50, no. 1, pp. 15169-15178, Jul. 2017, doi: 10.1016/j.ifacol.2017.08.2266.
- [Background] M. F. Penna et al., "Design and Administration of a Questionnaire for the User-Centered Design of a Novel Upper-Limb Assistive Device for Brachial Plexus Injury and Post-stroke Subjects," in Computers Helping People with Special Needs, K. Miesenberger, G. Kouroupetroglou, K. Mavrou, R. Manduchi, M. Covarrubias Rodriguez, and P. Penáz, Eds., in Lecture Notes in Computer Science. Cham: Springer International Publishing, 2022, pp. 420-427. doi: 10.1007/978-3-031-08645-8_49.
- [Background] Popovic MR, Thrasher TA, Zivanovic V, Takaki J, Hajek V. Neuroprosthesis for retraining reaching and grasping functions in severe hemiplegic patients. Neuromodulation. 2005 Jan;8(1):58-72. doi: 10.1111/j.1094-7159.2005.05221.x. PMID 22151384
- [Background] Resquin F, Cuesta Gomez A, Gonzalez-Vargas J, Brunetti F, Torricelli D, Molina Rueda F, Cano de la Cuerda R, Miangolarra JC, Pons JL. Hybrid robotic systems for upper limb rehabilitation after stroke: A review. Med Eng Phys. 2016 Nov;38(11):1279-1288. doi: 10.1016/j.medengphy.2016.09.001. Epub 2016 Sep 29. PMID 27692878
- [Background] Ferrante MA. Brachial plexopathies: classification, causes, and consequences. Muscle Nerve. 2004 Nov;30(5):547-68. doi: 10.1002/mus.20131. PMID 15452843